CLINICAL TRIAL: NCT01308697
Title: Operative Versus Non Operative Management of Flail Chest: A Randomized Controlled Feasibility Study
Brief Title: Flail Chest: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-03410
Record Dates: First submitted 2011-02-25; First posted 2011-03-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Flail Chest
Keywords: Flail; Chest
MeSH Terms: conditions — Flail Chest | interventions — Fracture Fixation, Internal; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative (Active Comparator): Operative intervention
  Interventions: Procedure: Operative fixation of flail chest
- Non Operative Treatment (Active Comparator): Non Operative management
  Interventions: Other: Non Operative management

INTERVENTIONS:
Procedure: Operative fixation of flail chest — Plate fixation
  Other Names: Internal Fixation
  Arms: Operative
Other: Non Operative management — Non Operative treatment of Flail Chest
  Other Names: Supportive care
  Arms: Non Operative Treatment

SUMMARY:
Flail chest refers to a section of the rib cage that has broken away from the surrounding ribs. Usually, more than one rib is involved, and they are broken in at least two places. Flail chest typically is the result of blunt chest trauma. As a result of flail chest, the chest wall becomes unstable and dangers of life threatening respiratory failure and hypoxemia (lack of oxygen to circulating blood which will lead to organ damage or failure)occur.

Currently, these injuries are treated non operatively. However, small case series have demonstrated that operative management can improve Intensive Care Unit (ICU) length of stay, improved pulmonary function and decreased pain leading to decreased duration of mechanical ventilation, and the incidence of complications related to this injury.

This study hopes to provide information on whether a prospective randomized trial is feasible by first undertaking a small pilot study to determine rate of recruitment, data collection methods, and integrity of study protocol.

Null Hypothesis 1: Enrollment of subjects with flail chest rib fractures into a prospective multi-centre RCT is not feasible and a larger clinical trial is unlikely to be completed.

DETAILED DESCRIPTION:
The optimum treatment of flail chest rib fractures is currently unknown. The standard of care for these injuries at most centers in North America, includes a progressive algorithm of epidural anesthesia, mechanical ventilation, and tracheostomy. Surgical management of flail chest injuries has previously been reserved for refractory cases unable to wean from mechanical ventilation or severe chest wall instability. However, the use of surgical stabilization of multiple rib fractures has demonstrated substantial improvements in ICU length of stay, duration of mechanical ventilation, and the incidences of pneumonia, tracheotomy, and reintubation. These results have been reported in small cases series without prospective or randomized trial designs.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years old
* greater than or equal to 4 adjacent rib fractures, with greater than one fracture per rib
* provide informed consent

Exclusion Criteria:

* Does not meet inclusion criteria
* Attending physician does not believe the subject will survive their injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Clinical outcomes | Day 1 Post Discharge
  Pilot study intends to review numerous clinical outcomes or variable of interest to assist in selecting a primary outcome and sample size for the future definitive trial. Currently Length of Stay in a high acuity unit is the planned primary outcome measure for the definitive trial

CONTACTS AND LOCATIONS:
Overall Officials: Peter J O'Brien, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia